CLINICAL TRIAL: NCT02763800
Title: Double-Blind, Randomised, Placebo-Controlled, Rising Multiple Dose Study to Investigate the Safety, Tolerability, Steady State Pharmacokinetic and Pharmacodynamic Profile of BIA 3-202, in Young Healthy Volunteers
Brief Title: Study to Investigate the Safety, Tolerability, Steady State Pharmacokinetic and Pharmacodynamic Profile of BIA 3-202
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-3202-02
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Nebicapone
MeSH Terms: conditions — Parkinson Disease | interventions — nebicapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: BIA 3-202 50 mg/placebo (Experimental): Group 1: BIA 3-202 50 mg/placebo on Day 1; BIA 3-202 50 mg/placebo b.i.d. on Days 3-8 inclusively; final single dose of BIA 3-202 50 mg/placebo on Day 9.
  50 mg BIA 3-202: 5 x 10 mg BIA 3-202 tablets
  Interventions: Drug: BIA 3-202; Drug: Placebo
- Group 2: BIA 3-202 100 mg/placebo (Experimental): Group 2: BIA 3-202 100 mg/placebo on Day 1; BIA 3-202 100 mg/placebo b.i.d. on Days 3-8 inclusively; final single dose of BIA 3-202 100 mg/placebo on Day 9.
  100 mg BIA 3-202: 1 x 100 mg BIA 3-202 tablet
  Interventions: Drug: BIA 3-202; Drug: Placebo
- Group 3: BIA 3-202 200 mg/placebo (Experimental): Group 3: BIA 3-202 200 mg/placebo on Day 1; BIA 3-202 200 mg/placebo b.i.d. on Days 3-8 inclusively; final single dose of BIA 3-202 200 mg/placebo on Day 9.
  200 mg BIA 3-202: 2 x 100 mg BIA 3-202 tablets
  Interventions: Drug: BIA 3-202; Drug: Placebo
- Group 4: BIA 3-202 200 mg/placebo (Experimental): Group 4: BIA 3-202 200 mg/placebo on Day 1; BIA 3-202 200 mg/placebo t.i.d. on Days 3-8 inclusively; final single dose of BIA 3-202 200 mg/placebo on Day 9.
  200 mg BIA 3-202: 2 x 100 mg BIA 3-202 tablets
  Interventions: Drug: BIA 3-202; Drug: Placebo

INTERVENTIONS:
Drug: BIA 3-202 — BIA 3-202 (50, 100 and 200 mg) was administered in the form of oral tablets, given with 200 ml potable water.
Drug: Placebo — Matched placebo was administered in the form of oral tablets, given with 200 ml potable water

SUMMARY:
The objectives as stated in the study protocol were as follows:

* To investigate the safety and tolerability of three multiple dose regimens of BIA 3-202 (50 mg twice a day, 100 mg twice a day and 200 mg twice a day in healthy young male volunteers). Part A
* To characterise the steady state pharmacokinetic and pharmacodynamic profile of BIA 3-202 in healthy young males. Part A
* To investigate the safety and tolerability of a single multiple dose regimen (dose to be determined from Part A) of BIA 3-202, in healthy elderly volunteers. Part B
* To characterise the steady state pharmacokinetic and pharmacodynamic profile of a single multiple dose regimen (dose to be determined from Part A) of BIA 3- 202 in healthy elderly volunteers. Part B

DETAILED DESCRIPTION:
This was designed as a single centre, phase I, double-blind, randomised, placebocontrolled study of three multiple rising doses in three sequential groups of 8 young male healthy volunteers (Part A) and a single group of healthy elderly volunteers (Part B).

In Part B, 12 healthy elderly volunteers were to be enrolled. Ten were to be randomly allocated to BIA 3-202 and two to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 18-35 years, with a body mass index (BMI) of 19-28 kg/m2.
* Subjects who were healthy as determined by pre-study medical history, physical examination and 12-lead ECG.
* Subjects who had clinical laboratory tests acceptable to the investigator.
* Subjects who were negative for HbsAg, anti-HCV and HIV I and II tests at screening.
* Subjects who were negative for drugs of abuse and alcohol tests at screening and admission.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism.
* Subjects who had a history of drug abuse.
* Subjects who consumed more than 28 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn).
* Subjects who had an acute infection such as influenza at the time of screening and/or admission.
* Subjects who had used prescription drugs within 4 weeks of first dosing.
* Subjects who had used over the counter medication, excluding routine vitamins but including mega dose vitamin therapy, within one week of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 3 months of their first admission to this study.
* Subjects who had previously received BIA 3-202.
* Subjects who had donated and/or received any blood or blood products within 3 months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2000-09; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) - D1 | Day 1
Time of maximum observed concentration (tmax) - D1 | Day 1
Area under the plasma concentration time curve to last measurable time point (AUC0-t) - D1 | Day 1
Area under the plasma concentration time curve extrapolated to infinity (AUC0-∞) - D1 | Day 1
Maximum observed plasma concentration (Cmax) - D9 | Day 9
Time of maximum observed concentration (tmax) - D9 | Day 9
Area under the plasma concentration time curve to last measurable time point (AUC0-t) - D9 | Day 9
Area under the plasma concentration time curve extrapolated to infinity (AUC0-∞) - D9 | Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's Drug Research Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No